CLINICAL TRIAL: NCT00531284
Title: Phase 1b/2, Multicenter Open-label Study of the Safety and Activity of Carfilzomib in Subjects With Relapsed Solid Tumors, Multiple Myeloma or Lymphoma
Brief Title: Phase 1b/2 Study of Carfilzomib in Relapsed Solid Tumors, Multiple Myeloma, or Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PX-171-007
Record Dates: First submitted 2007-09-14; First posted 2007-09-18 (Estimated); Results first posted 2015-12-09 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-07

CONDITIONS: Ovarian Cancer; Renal Cancer; Non-small Cell Lung Cancer; Small Cell Lung Cancer; Solid Tumors; Multiple Myeloma; Lymphoma
Keywords: Non-small cell lung carcinoma; Small-cell lung carcinoma; Ovarian Cancer; Renal Cancer; Other solid tumors; multiple myeloma; lymphoma
MeSH Terms: conditions — Ovarian Neoplasms; Kidney Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Multiple Myeloma; Lymphoma | interventions — carfilzomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (17):
- Phase 1B Solid Tumors: Carfilzomib 20 mg/m² Bolus (Experimental): Participants received carfilzomib 20 mg/m² administered by bolus intravenous infusion over 2-10 minutes on Days 1, 2, 8, 9, 15, and 16 of a 28-day cycle. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
  Interventions: Drug: Carfilzomib
- Phase 1B Solid Tumors: Carfilzomib 20/27 mg/m² Bolus (Experimental): Participants received carfilzomib 20 mg/m² administered by bolus intravenous infusion over 2-10 minutes on Cycle 1 Days 1 and 2 only, then 27 mg/m² on Days 8, 9, 15 and 16 and thereafter for the remainder of treatment. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
  Interventions: Drug: Carfilzomib
- Phase 1B Solid Tumors: Carfilzomib 20/36 mg/m² Bolus (Experimental): Participants received carfilzomib 20 mg/m² administered by bolus intravenous infusion over 2-10 minutes on Cycle 1 Days 1 and 2 only, then 36 mg/m² on Days 8, 9, 15 and 16 and thereafter for the remainder of treatment. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
  Interventions: Drug: Carfilzomib
- Phase 2 Solid Tumors: Carfilzomib 20/36 mg/m² Bolus (Experimental): Participants received carfilzomib 20 mg/m² administered by bolus intravenous infusion over 2-10 minutes on Cycle 1 Days 1 and 2 only, then 36 mg/m² on Days 8, 9, 15 and 16 and thereafter for the remainder of treatment. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
  Interventions: Drug: Carfilzomib
- Phase 1B Solid Tumors: Carfilzomib 36 mg/m² (Experimental): Participants received carfilzomib 36 mg/m² administered by intravenous infusion over 30 minutes on Days 1, 2, 8, 9, 15, and 16 of a 28-day cycle for at least 2 cycles. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
  Interventions: Drug: Carfilzomib
- Phase 1B Solid Tumors: Carfilzomib 45 mg/m² (Experimental): Participants received carfilzomib 45 mg/m² administered by intravenous infusion over 30 minutes on Days 1, 2, 8, 9, 15, and 16 of a 28-day cycle for at least 2 cycles. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
  Interventions: Drug: Carfilzomib
- Phase 1B Solid Tumors: Carfilzomib 20/45 mg/m² (Experimental): Participants received carfilzomib 20 mg/m² administered by intravenous infusion over 30 minutes on Cycle 1 Days 1 and 2 only, then 45 mg/m² on Days 8, 9, 15 and 16 and thereafter for the remainder of treatment. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
  Interventions: Drug: Carfilzomib
- Phase 1B Solid Tumors: Carfilzomib 20/56 mg/m² (Experimental): Participants received carfilzomib 20 mg/m² administered by intravenous infusion over 30 minutes on Cycle 1 Days 1 and 2 only, then 56 mg/m² on Days 8, 9, 15 and 16 and thereafter for the remainder of treatment. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
  Interventions: Drug: Carfilzomib
- Phase 1B Solid Tumors: Carfilzomib 20/70 mg/m² (Experimental): Participants received carfilzomib 20 mg/m² administered by intravenous infusion over 30 minutes on Cycle 1 Days 1 and 2 only, then 70 mg/m² on Days 8, 9, 15 and 16 and thereafter for the remainder of treatment. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
  Interventions: Drug: Carfilzomib
- Phase 1b Multiple Myeloma: Carfilzomib 20/36 mg/m² (Experimental): Participants received carfilzomib 20 mg/m² administered by intravenous infusion over 30 minutes on Cycle 1 Days 1 and 2 only, then 36 mg/m² on Days 8, 9, 15 and 16 and thereafter for the remainder of treatment. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
  Interventions: Drug: Carfilzomib
- Phase 1b Multiple Myeloma: Carfilzomib 20/45 mg/m² (Experimental): Participants received carfilzomib 20 mg/m² administered by intravenous infusion over 30 minutes on Cycle 1 Days 1 and 2 only, then 45 mg/m² on Days 8, 9, 15 and 16 and thereafter for the remainder of treatment. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
  Interventions: Drug: Carfilzomib
- Phase 1b Multiple Myeloma: Carfilzomib 20/56 mg/m² (Experimental): Participants received carfilzomib 20 mg/m² administered by intravenous infusion over 30 minutes on Cycle 1 Days 1 and 2 only, then 56 mg/m² on Days 8, 9, 15 and 16 and thereafter for the remainder of treatment. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
  Interventions: Drug: Carfilzomib
- Phase 1b Multiple Myeloma: Carfilzomib 20/70 mg/m² (Experimental): Participants received carfilzomib 20 mg/m² administered by intravenous infusion over 30 minutes on Cycle 1 Days 1 and 2 only, then 70 mg/m² on Days 8, 9, 15 and 16 and thereafter for the remainder of treatment. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
  Interventions: Drug: Carfilzomib
- Phase 1b Lymphoma: Carfilzomib 20/56 mg/m² (Experimental): Participants received carfilzomib 20 mg/m² administered by intravenous infusion over 30 minutes on Cycle 1 Days 1 and 2 only, then 56 mg/m² on Days 8, 9, 15 and 16 and thereafter for the remainder of treatment. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
  Interventions: Drug: Carfilzomib
- Phase 1b Lymphoma: Carfilzomib 20/70 mg/m² (Experimental): Participants received carfilzomib 20 mg/m² administered by intravenous infusion over 30 minutes on Cycle 1 Days 1 and 2 only, then 70 mg/m² on Days 8, 9, 15 and 16 and thereafter for the remainder of treatment. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
  Interventions: Drug: Carfilzomib
- Phase 1b MM: Carfilzomib 20/45 mg/m² + Dexamethasone (Experimental): Participants received carfilzomib 20 mg/m² administered by intravenous infusion over 30 minutes on Cycle 1 Days 1 and 2 only, then 45 mg/m² on Days 8, 9, 15 and 16 and thereafter for the remainder of treatment plus dexamethasone 40 mg weekly. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone
- Phase 1b MM: Carfilzomib 20/56 mg/m² + Dexamethasone (Experimental): Participants received carfilzomib 20 mg/m² administered by intravenous infusion over 30 minutes on Cycle 1 Days 1 and 2 only, then 56 mg/m² on Days 8, 9, 15 and 16 and thereafter for the remainder of treatment plus dexamethasone 40 mg weekly. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib — Administered by intravenous (IV) bolus (2-10 minute) infusion or 30 minute infusion
  Other Names: Kyprolis
Drug: Dexamethasone — Administered orally or by IV infusion prior to carfilzomib
  Arms: Phase 1b MM: Carfilzomib 20/45 mg/m² + Dexamethasone; Phase 1b MM: Carfilzomib 20/56 mg/m² + Dexamethasone

SUMMARY:
The primary objectives of this Phase 1b/2 study were as follows:

* Phase 1b (Bolus and Infusion): To evaluate the safety and tolerability of carfilzomib in patients with relapsed solid tumors and in patients with relapsed and/or refractory multiple myeloma and in patients with refractory lymphoma.
* Phase 2 (Bolus): To evaluate the overall response rate (ORR) after 4 cycles of carfilzomib in patients with relapsed solid tumors.

ELIGIBILITY:
Inclusion Criteria:

Disease related

Phase 1 Subjects (Bolus and Infusion):

Solid Tumor:

* Histologically confirmed advanced solid tumor
* 1 to 3 prior treatment regimens
* At least one site of radiographically measurable disease of ≥ 2 cm in the largest dimension by traditional computed tomography (CT) scanning technique or ≥ 1 cm in the largest dimension by spiral CT scanning (per Response Evaluation Criteria in Solid Tumors [RECIST] criteria); or if, in the Principal Investigator's opinion, evaluable disease can be reliably and consistently followed, the subject may be eligible upon approval by the Medical Monitor

Multiple Myeloma (MM):

* Relapsed and/or refractory multiple myeloma following 2 or more prior treatment regimens.
* Measurable disease as indicated by one or more of the following:
* Serum M-protein ≥ 1 g/dL
* Urine M-protein ≥ 200 mg/24 hr
* Serum Free Light Chain: Involved free light chain (FLC) level ≥ 10 mg/dL provided serum FLC ratio is abnormal

Lymphoma:

* Histologically or cytologically confirmed lymphoma.
* Patients must have had an initial diagnosis of indolent non-Hodgkin lymphoma (NHL) (including follicular, small lymphocytic, lymphoplasmacytoid, and marginal zone lymphoma), indolent disease that transformed to a more aggressive subtype, as previously described or patients may have mantle cell lymphoma.
* Patients are required to have received prior rituximab (alone or combined with other treatment) and are considered refractory to (defined as no response, or progression within 6 months of completing therapy) or intolerant of continued rituximab.
* Patients may have received up to a maximum of four prior unique chemotherapy regimens, including if not contra-indicated autologous stem-cell transplantation (ASCT).
* For patients to enroll in the expanded dose group for lymphoma, patients must have measurable disease

Phase 2 Bolus Subjects:

-Histologically confirmed advanced solid tumor diagnosis and:

* Non-small cell lung cancer (NSCLC): Failed at least 1 prior platinum-based chemotherapy regimen but not more than 3 prior therapies for metastatic disease
* Small cell lung cancer (SCLC): Failed 1 to 3 prior chemotherapy regimens
* Ovarian: Failed at least 1 prior platinum-based chemotherapy regimen but not more than 4 therapies for metastatic disease
* Renal: Failed at least 2 prior chemotherapy regimens for metastatic disease
* Other solid tumor types: Failed at least 1 prior chemotherapy regimen for metastatic or relapsed disease and for which standard of care therapy is no longer effective or does not exist
* At least one site of radiographically measurable disease of ≥ 2 cm in the largest dimension by traditional CT scanning technique or ≥ 1 cm in the largest dimension by spiral CT scanning (per RECIST criteria); or if, in the Principal Investigator's opinion, evaluable disease can be reliably and consistently followed, the subject may be eligible upon approval by the Medical Monitor

Demographic

* Males and females ≥ 18 years of age
* Life expectancy of more than 3 months
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2

Laboratory

* Adequate hepatic function, with bilirubin 1.5 times the upper limit of normal (ULN), and alanine aminotransferase (ALT) 3 times ULN
* Absolute neutrophil count (ANC) > 1000/mm³, hemoglobin ≥ 8 gm/dL for solid tumors or 7.0 gm/dL for MM, and platelet count ≥ 100,000/mm³ for solid tumors or ≥ 30,000/mm³ for MM.

  * Subjects should not have received platelet transfusions for at least 1 week prior to screening
  * Screening ANC should be independent of granulocyte- and granulocyte/macrophage colony stimulating factor (G-CSF and GM-CSF) support for at least 1 week and of pegylated G-CSF for ≥ 2 weeks
  * Subjects may receive red blood cell (RBC) transfusions or receive supportive care with erythropoietin or darbepoetin in accordance with institutional guidelines
* Calculated or measured creatinine clearance (CrCl) of ≥ 20 mL/minute calculated using the formula of Cockcroft and Gault. Subjects with calculated CrCl < 20 mL/min may be allowed, only with prior approval by the Medical Monitor.

Ethical/Other

* Written informed consent in accordance with federal, local, and institutional guidelines
* Female subjects of childbearing potential must have a negative serum or urine pregnancy test within 3 days of the first dose and agree to use dual methods of contraception during the study and for 3 months following the last dose of study drug. Post-menopausal females (> 45 years old and without menses for > 1 year) and surgically sterilized females are exempt from these requirements. Male subjects must use an effective barrier method of contraception during the study and for 3 months following the last dose if sexually active with a female of childbearing potential.

Exclusion Criteria:

Disease Related

* Chemotherapy with approved or investigational anticancer therapeutics, including steroid therapy, within 3 weeks prior to first dose or 6 weeks for antibody therapy
* Radiation therapy or immunotherapy within 3 weeks prior to first dose (except for antibody therapy, where 6 weeks is required); localized radiation therapy within 1 week prior to first dose
* Subjects with prior brain metastases are permitted, but must have completed treatment and have no evidence of active central nervous system (CNS) disease for at least 4 weeks prior to first dose
* For lymphoma patients; patients with prior stem cell transplant therapy (autologous SCT within the prior 8 weeks; allogeneic SCT within the prior 16 weeks). Patients with prior allogeneic SCT should not have evidence of moderate-to-severe graft-versus-host disease (GVHD)
* Evidence of CNS lymphoma
* Participation in an investigational therapeutic study within 3 weeks prior to first dose
* Prior treatment with carfilzomib

Concurrent Conditions

* Major surgery within 3 weeks prior to first dose
* Congestive heart failure (New York Heart Association class III to IV), symptomatic ischemia, conduction abnormalities uncontrolled by conventional intervention, or myocardial infarction within 3 months prior to first dose
* Acute active infection requiring systemic antibiotics, antivirals, or antifungals within 2 weeks prior to first dose
* Known or suspected human immunodeficiency virus (HIV) infection or subjects who are HIV seropositive
* Active hepatitis A, B, or C infection
* Significant neuropathy (Grade 3, Grade 4, or Grade 2 with pain) at the time of the first dose
* Subjects with pleural effusions requiring routine thoracentesis or ascites requiring routine paracentesis
* Subjects at risk* in whom the required program of oral and intravenous fluid hydration is contraindicated, e.g., due to pre-existing pulmonary, cardiac, or renal impairment

  * High risk for Tumor Lysis Syndrome.

Ethical / Other

* Female subjects who are pregnant or lactating
* Any clinically significant psychiatric or medical condition that in the opinion of the Investigator could interfere with protocol adherence or a subject's ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2007-09; Primary Completion 2014-10 (Actual); Study Completion 2017-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (7):
- United States (7):
  - Pinnacle Oncology, Scottsdale, Arizona
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Northwestern University, Chicago, Illinois
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas

REFERENCES:
- [Derived] Papadopoulos KP, Siegel DS, Vesole DH, Lee P, Rosen ST, Zojwalla N, Holahan JR, Lee S, Wang Z, Badros A. Phase I study of 30-minute infusion of carfilzomib as single agent or in combination with low-dose dexamethasone in patients with relapsed and/or refractory multiple myeloma. J Clin Oncol. 2015 Mar 1;33(7):732-9. doi: 10.1200/JCO.2013.52.3522. Epub 2014 Sep 15. PMID 25225420
- [Derived] Ohshima-Hosoyama S, Davare MA, Hosoyama T, Nelon LD, Keller C. Bortezomib stabilizes NOXA and triggers ROS-associated apoptosis in medulloblastoma. J Neurooncol. 2011 Dec;105(3):475-83. doi: 10.1007/s11060-011-0619-0. Epub 2011 Jun 3. PMID 21633906

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with relapsed solid tumors (non-small and small cell lung, ovarian, renal, any other solid tumor type), multiple myeloma or lymphoma were enrolled at 7 sites in the US.
  Under the original protocol patients received a bolus intravenous (IV) infusion of carfilzomib; patients enrolled under Amendments 2 to 4 received a 30-minute IV infusion.
Pre-assignment Details: Phase 1b followed a 3+3 dose-escalation design to determine the maximum tolerated dose (MTD). For Phase 2 (bolus), a Simon 2-stage design was planned using the MTD from phase 1b. The first stage of the Simon's 2-stage design was carried out; however, the study did not progress to the second stage.
Groups:
- P1B ST: CFZ 20 mg/m² Bolus: Participants with solid tumors (ST) received carfilzomib (CFZ) 20 mg/m² administered by bolus intravenous infusion over 2-10 minutes on Days 1, 2, 8, 9, 15, and 16 of a 28-day cycle. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
- P1B ST: CFZ 20/27 mg/m² Bolus: Participants with solid tumors received carfilzomib 20 mg/m² administered by bolus intravenous infusion over 2-10 minutes on Cycle 1 Days 1 and 2 only, then 27 mg/m² on Days 8, 9, 15 and 16 and thereafter for the remainder of treatment. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
- P1B ST: CFZ 20/36 mg/m² Bolus; P2 ST: CFZ 20/36 mg/m² Bolus: Participants with solid tumors received carfilzomib 20 mg/m² administered by bolus intravenous infusion over 2-10 minutes on Cycle 1 Days 1 and 2 only, then 36 mg/m² on Days 8, 9, 15 and 16 and thereafter for the remainder of treatment. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
- P1B ST: CFZ 36 mg/m²: Participants with solid tumors received carfilzomib 36 mg/m² administered by intravenous infusion over 30 minutes on Days 1, 2, 8, 9, 15, and 16 of a 28-day cycle for at least 2 cycles. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
- P1B ST: CFZ 45 mg/m²: Participants with solid tumors received carfilzomib 45 mg/m² administered by intravenous infusion over 30 minutes on Days 1, 2, 8, 9, 15, and 16 of a 28-day cycle for at least 2 cycles. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
- P1B ST: CFZ 20/45 mg/m²: Participants with solid tumors received carfilzomib 20 mg/m² administered by intravenous infusion over 30 minutes on Cycle 1 Days 1 and 2 only, then 45 mg/m² on Days 8, 9, 15 and 16 and thereafter for the remainder of treatment. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
- P1B ST: CFZ 20/56 mg/m²: Participants with solid tumors received carfilzomib 20 mg/m² administered by intravenous infusion over 30 minutes on Cycle 1 Days 1 and 2 only, then 56 mg/m² on Days 8, 9, 15 and 16 and thereafter for the remainder of treatment. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
- P1B ST: CFZ 20/70 mg/m²: Participants with solid tumors received carfilzomib 20 mg/m² administered by intravenous infusion over 30 minutes on Cycle 1 Days 1 and 2 only, then 70 mg/m² on Days 8, 9, 15 and 16 and thereafter for the remainder of treatment. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
- P1B MM: CFZ 20/36 mg/m²: Participants with multiple myeloma received carfilzomib 20 mg/m² administered by intravenous infusion over 30 minutes on Cycle 1 Days 1 and 2 only, then 36 mg/m² on Days 8, 9, 15 and 16 and thereafter for the remainder of treatment. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
- P1B MM: CFZ 20/45 mg/m²: Participants with multiple myeloma (MM) received carfilzomib 20 mg/m² administered by intravenous infusion over 30 minutes on Cycle 1 Days 1 and 2 only, then 45 mg/m² on Days 8, 9, 15 and 16 and thereafter for the remainder of treatment. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
- P1b MM: CFZ 20/56 mg/m²: Participants with multiple myeloma received carfilzomib 20 mg/m² administered by intravenous infusion over 30 minutes on Cycle 1 Days 1 and 2 only, then 56 mg/m² on Days 8, 9, 15 and 16 and thereafter for the remainder of treatment. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
- P1B MM: CFZ 20/70 mg/m²: Participants with multiple myeloma received carfilzomib 20 mg/m² administered by intravenous infusion over 30 minutes on Cycle 1 Days 1 and 2 only, then 70 mg/m² on Days 8, 9, 15 and 16 and thereafter for the remainder of treatment. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
- P1B LYM: CFZ 20/56 mg/m²: Participants with lymphoma (LYM) received carfilzomib 20 mg/m² administered by intravenous infusion over 30 minutes on Cycle 1 Days 1 and 2 only, then 56 mg/m² on Days 8, 9, 15 and 16 and thereafter for the remainder of treatment. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
- P1B LYM: CFZ 20/70 mg/m²: Participants with lymphoma received carfilzomib 20 mg/m² administered by intravenous infusion over 30 minutes on Cycle 1 Days 1 and 2 only, then 70 mg/m² on Days 8, 9, 15 and 16 and thereafter for the remainder of treatment. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
- P1B MM: CFZ 20/45 mg/m² + Dex: Participants with multiple myeloma received carfilzomib 20 mg/m² administered by intravenous infusion over 30 minutes on Cycle 1 Days 1 and 2 only, then 45 mg/m² on Days 8, 9, 15 and 16 and thereafter for the remainder of treatment plus dexamethasone 40 mg weekly. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
- P1B MM: CFZ 20/56 mg/m² + Dex: Participants with multiple myeloma received carfilzomib 20 mg/m² administered by intravenous infusion over 30 minutes on Cycle 1 Days 1 and 2 only, then 56 mg/m² on Days 8, 9, 15 and 16 and thereafter for the remainder of treatment plus dexamethasone 40 mg weekly. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
Period: Overall Study
Arm/Group | P1B ST: CFZ 20 mg/m² Bolus | P1B ST: CFZ 20/27 mg/m² Bolus | P1B ST: CFZ 20/36 mg/m² Bolus | P2 ST: CFZ 20/36 mg/m² Bolus | P1B ST: CFZ 36 mg/m² | P1B ST: CFZ 45 mg/m² | P1B ST: CFZ 20/45 mg/m² | P1B ST: CFZ 20/56 mg/m² | P1B ST: CFZ 20/70 mg/m² | P1B MM: CFZ 20/36 mg/m² | P1B MM: CFZ 20/45 mg/m² | P1b MM: CFZ 20/56 mg/m² | P1B MM: CFZ 20/70 mg/m² | P1B LYM: CFZ 20/56 mg/m² | P1B LYM: CFZ 20/70 mg/m² | P1B MM: CFZ 20/45 mg/m² + Dex | P1B MM: CFZ 20/56 mg/m² + Dex
Started | 3 | 4 | 7 | 65 | 6 | 7 | 6 | 10 | 11 | 4 | 3 | 24 | 2 | 3 | 7 | 14 | 8
Completed | 0 (Indicates participants who completed 12 cycles of study drug) | 0 (Indicates participants who completed 12 cycles of study drug) | 1 (Indicates participants who completed 12 cycles of study drug) | 2 (Indicates participants who completed 12 cycles of study drug) | 0 (Indicates participants receiving treatment as of the data cut-off date of 07 October 2014) | 0 (Indicates participants receiving treatment as of the data cut-off date of 07 October 2014) | 0 (Indicates participants receiving treatment as of the data cut-off date of 07 October 2014) | 0 (Indicates participants receiving treatment as of the data cut-off date of 07 October 2014) | 0 (Indicates participants receiving treatment as of the data cut-off date of 07 October 2014) | 0 (Indicates participants receiving treatment as of the data cut-off date of 07 October 2014) | 0 (Indicates participants receiving treatment as of the data cut-off date of 07 October 2014) | 0 (Indicates participants receiving treatment as of the data cut-off date of 07 October 2014) | 0 (Indicates participants receiving treatment as of the data cut-off date of 07 October 2014) | 0 (Indicates participants receiving treatment as of the data cut-off date of 07 October 2014) | 3 (Indicates participants receiving treatment as of the data cut-off date of 07 October 2014) | 2 (Indicates participants receiving treatment as of the data cut-off date of 07 October 2014) | 0 (Indicates participants receiving treatment as of the data cut-off date of 07 October 2014)
Not Completed | 3 | 4 | 6 | 63 | 6 | 7 | 6 | 10 | 11 | 4 | 3 | 24 | 2 | 3 | 4 | 12 | 8
Not completed — Progressive Disease | 1 | 3 | 5 | 42 | 4 | 4 | 3 | 8 | 6 | 3 | 3 | 14 | 2 | 1 | 2 | 11 | 5
Not completed — Adverse Event | 0 | 1 | 1 | 7 | 0 | 2 | 3 | 2 | 3 | 0 | 0 | 5 | 0 | 1 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 1 | 1
Not completed — Other | 1 | 0 | 0 | 10 | 2 | 1 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | P1B ST: CFZ 20 mg/m² Bolus | P1B ST: CFZ 20/27 mg/m² Bolus | P1B ST: CFZ 20/36 mg/m² Bolus | P2 ST: CFZ 20/36 mg/m² Bolus | P1B ST: CFZ 36 mg/m² | P1B ST: CFZ 45 mg/m² | P1B ST: CFZ 20/45 mg/m² | P1B ST: CFZ 20/56 mg/m² | P1B ST: CFZ 20/70 mg/m² | P1B MM: CFZ 20/36 mg/m² | P1B MM: CFZ 20/45 mg/m² | P1b MM: CFZ 20/56 mg/m² | P1B MM: CFZ 20/70 mg/m² | P1B LYM: CFZ 20/56 mg/m² | P1B LYM: CFZ 20/70 mg/m² | P1B MM: CFZ 20/45 mg/m² + Dex | P1B MM: CFZ 20/56 mg/m² + Dex | Total
Number analyzed (Participants) | 3 | 4 | 7 | 65 | 6 | 7 | 6 | 10 | 11 | 4 | 3 | 24 | 2 | 3 | 7 | 14 | 8 | 184
Age, Continuous [Mean (Standard Deviation); unit: years]
  Bolus Groups | 47.3 (14.74) | 60.8 (8.81) | 60.0 (11.72) | 62.0 (9.97) | NA (NA) — Not applicable for infusion arms | NA (NA) — Not applicable for infusion arms | NA (NA) — Not applicable for infusion arms | NA (NA) — Not applicable for infusion arms | NA (NA) — Not applicable for infusion arms | NA (NA) — Not applicable for infusion arms | NA (NA) — Not applicable for infusion arms | NA (NA) — Not applicable for infusion arms | NA (NA) — Not applicable for infusion arms | NA (NA) — Not applicable for infusion arms | NA (NA) — Not applicable for infusion arms | NA (NA) — Not applicable for infusion arms | NA (NA) — Not applicable for infusion arms | 62.20 (10.43)
  30-minute Infusion Groups | NA (NA) — Not applicable for bolus arms | NA (NA) — Not applicable for bolus arms | NA (NA) — Not applicable for bolus arms | NA (NA) — Not applicable for bolus arms | 60.0 (5.18) | 69.9 (11.10) | 61.2 (10.38) | 61.4 (7.40) | 61.6 (11.58) | 63.3 (3.77) | 72.0 (5.57) | 62.7 (9.88) | 69.5 (12.02) | 58.7 (10.69) | 65.4 (10.31) | 58.6 (9.54) | 58.3 (6.14) | 62.3 (9.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 4 | 38 | 0 | 4 | 3 | 5 | 4 | 2 | 1 | 7 | 1 | 1 | 3 | 4 | 1 | 80
  Male | 2 | 3 | 3 | 27 | 6 | 3 | 3 | 5 | 7 | 2 | 2 | 17 | 1 | 2 | 4 | 10 | 7 | 104
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Scale used to assess how a patient's disease is progressing, how the disease affects the daily living abilities of the patient: 0 = Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity, ambulatory, able to carry out work of a light nature; 2 = Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about > 50% of waking hours; 3 = Capable of only limited self care, confined to a bed or chair > 50% of waking hours; 4 = Completely disabled, confined to bed or chair; 5 = Dead.
  participants
    0 | 1 | 3 | 4 | 27 | 2 | 1 | 0 | 2 | 4 | 4 | 0 | 8 | 0 | 2 | 3 | 7 | 5 | 73
    1 | 2 | 1 | 3 | 35 | 4 | 4 | 6 | 7 | 7 | 0 | 2 | 15 | 1 | 0 | 3 | 6 | 3 | 99
    2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 9
    Missing | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants With Dose-limiting Toxicities (DLT)
Description: Participants were evaluated for dose-limiting toxicities according to the Common Terminology Criteria for Adverse Events (CTCAE) of the National Cancer Institute (NCI) version 3.0.
  A DLT was defined as treatment-related ≥ Grade 2 neuropathy with pain, ≥ Grade 3 non-hematologic toxicity, Grade 4 neutropenia or thrombocytopenia lasting 7 or more days, or thrombocytopenia with bleeding.
  The maximum tolerated dose (MTD) for each of the 3 populations (solid tumor, multiple myeloma, and lymphoma) was defined as the dose level at which < 33% of participants experienced a dose-limiting toxicity during the first 28-day cycle.
Time Frame: 28 days
Population: Dose-limiting toxicity analysis was based on subsets of the safety population including participants exposed to carfilzomib in Cycle 1 who experienced a DLT or completed 28 days of evaluation after the first dose of carfilzomib. Participants enrolled into the expansion cohorts (MTD dose expansion, carfilzomib + DEX) were not evaluated for DLT.
Measure: Number; unit: participants
Arm/Group | P1B ST: CFZ 20 mg/m² Bolus | P1B ST: CFZ 20/27 mg/m² Bolus | P1B ST: CFZ 20/36 mg/m² Bolus | P1B ST: CFZ 36 mg/m² | P1B ST: CFZ 45 mg/m² | P1B ST: CFZ 20/45 mg/m² | P1B ST: CFZ 20/56 mg/m² | P1B ST: CFZ 20/70 mg/m² | P1B MM: CFZ 20/36 mg/m² | P1B MM: CFZ 20/45 mg/m² | P1b MM: CFZ 20/56 mg/m² | P1B MM: CFZ 20/70 mg/m² | P1B LYM: CFZ 20/56 mg/m² | P1B LYM: CFZ 20/70 mg/m²
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 6 | 6 | 3 | 6 | 4 | 3 | 6 | 2 | 3 | 7
participants | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 1

2. Primary Outcome: Phase 2: Percentage of Participants With an Overall Response After 4 Treatment Cycles
Description: Overall response is defined as participants with a best overall response of complete response (CR), partial response (PR) or stable disease (SD) after 4 cycles, assessed by the Investigator using tumor measurement and according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
  CR: Disappearance of all target and non-target lesions and no new lesions;
  PR: Disappearance of all target lesions, persistence of one or more non-target lesion(s) or/and maintenance of tumor marker level above the normal limits and no lesions, or, at least a 30% decrease in the size of target lesions and no progression of existing non-target lesions or any new lesions.
  SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest size since the treatment started, and no progression of existing non-target lesions or any new lesions.
Time Frame: 4 months
Population: Phase 2 Safety population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- P2 ST: CFZ 20/36 mg/m² Bolus: Participants with solid tumors received carfilzomib 20 mg/m² administered by bolus intravenous infusion over 2-10 minutes on Cycle 1 Days 1 and 2 only, then 36 mg/m² on Days 8, 9, 15 and 16 and thereafter for the remainder of treatment.
Arm/Group | P2 ST: CFZ 20/36 mg/m² Bolus
Number analyzed (Participants) | 65
percentage of participants | 15.4 [7.6 to 26.5]

3. Secondary Outcome: Percentage of Participants With an Overall Response Throughout the Study
Description: Solid tumor participants were evaluated for disease response according to RECIST, Version 1.1. Multiple myeloma participants were evaluated using the International Myeloma Working Group (IMWG) Uniform Response Criteria with the addition of minimal response (MR) based on the European Group for Blood and Marrow Transplant Group (EBMT). Non-Hodgkin lymphoma (NHL) participants were evaluated using the International Workshop NHL criteria. Waldenström macroglobulinemia (WM) participants were evaluated using Criteria from the Sixth International Workshop for WM.
  Overall response is defined in Outcome Measure 2 for participants with solid tumors. For NHL, overall response is defined as a best overall response of CR or PR. For multiple myeloma and WM, overall response is defined as participants with a best overall response of stringent complete response (sCR), CR, very good partial response (VGPR) or PR.
Time Frame: Tumor assessments occurred at the end of Cycle 2, 4, 6, 9, and 12 and continued every 3 cycles thereafter up to 6 months after last dose. Analysis includes data up to the data cut-off date of 07 October 2014; maximum duration of treatment was 35 months.
Population: Safety Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- P1B NHL: CFZ 20/56 mg/m²: Participants with non-Hodgkin's lymphoma (NHL) received carfilzomib 20 mg/m² administered by intravenous infusion over 30 minutes on Cycle 1 Days 1 and 2 only, then 56 mg/m² on Days 8, 9, 15 and 16 and thereafter for the remainder of treatment. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
- P1B NHL: CFZ 20/70 mg/m²: Participants with non-Hodgkin's lymphoma received carfilzomib 20 mg/m² administered by intravenous infusion over 30 minutes on Cycle 1 Days 1 and 2 only, then 70 mg/m² on Days 8, 9, 15 and 16 and thereafter for the remainder of treatment. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
- P1B WM: CFZ 20/56 mg/m²: Participants with Waldenstrom macroglobulinemia (WM) received carfilzomib 20 mg/m² administered by intravenous infusion over 30 minutes on Cycle 1 Days 1 and 2 only, then 56 mg/m² on Days 8, 9, 15 and 16 and thereafter for the remainder of treatment. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
- P1B WM: CFZ 20/70 mg/m²: Participants with Waldenstrom macroglobulinemia (WM) received carfilzomib 20 mg/m² administered by intravenous infusion over 30 minutes on Cycle 1 Days 1 and 2 only, then 70 mg/m² on Days 8, 9, 15 and 16 and thereafter for the remainder of treatment. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
Arm/Group | P1B ST: CFZ 20 mg/m² Bolus | P1B ST: CFZ 20/27 mg/m² Bolus | P1B ST: CFZ 20/36 mg/m² Bolus | P2 ST: CFZ 20/36 mg/m² Bolus | P1B ST: CFZ 36 mg/m² | P1B ST: CFZ 45 mg/m² | P1B ST: CFZ 20/45 mg/m² | P1B ST: CFZ 20/56 mg/m² | P1B ST: CFZ 20/70 mg/m² | P1B MM: CFZ 20/36 mg/m² | P1B MM: CFZ 20/45 mg/m² | P1b MM: CFZ 20/56 mg/m² | P1B MM: CFZ 20/70 mg/m² | P1B NHL: CFZ 20/56 mg/m² | P1B NHL: CFZ 20/70 mg/m² | P1B WM: CFZ 20/56 mg/m² | P1B WM: CFZ 20/70 mg/m² | P1B MM: CFZ 20/45 mg/m² + Dex | P1B MM: CFZ 20/56 mg/m² + Dex
Number analyzed (Participants) | 3 | 4 | 7 | 65 | 6 | 7 | 6 | 10 | 11 | 4 | 3 | 24 | 2 | 2 | 3 | 1 | 4 | 14 | 8
percentage of participants | 100.0 [29.2 to 100.0] | 0.0 [0.0 to 60.2] | 42.9 [9.9 to 81.6] | 38.5 [26.7 to 51.4] | 33.3 [4.3 to 77.7] | 28.6 [3.7 to 71.0] | 50.0 [11.8 to 88.2] | 10.0 [0.3 to 44.5] | 36.4 [10.9 to 69.2] | 50.0 [6.8 to 93.2] | 33.3 [0.8 to 90.6] | 50.0 [29.1 to 70.9] | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 100.0 [2.5 to 100.0] | 100.0 [39.8 to 100.0] | 64.3 [35.1 to 87.2] | 37.5 [8.5 to 75.5]

4. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time from first evidence of a partial response or better (the first observation of PR before confirmation) to disease progression, with deaths owing to causes other than progression censored.
Time Frame: as for outcome 3
Population: Safety Population with a partial response or better
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | P1B ST: CFZ 20 mg/m² Bolus | P1B ST: CFZ 20/27 mg/m² Bolus | P1B ST: CFZ 20/36 mg/m² Bolus | P2 ST: CFZ 20/36 mg/m² Bolus | P1B ST: CFZ 36 mg/m² | P1B ST: CFZ 45 mg/m² | P1B ST: CFZ 20/45 mg/m² | P1B ST: CFZ 20/56 mg/m² | P1B ST: CFZ 20/70 mg/m² | P1B MM: CFZ 20/36 mg/m² | P1B MM: CFZ 20/45 mg/m² | P1b MM: CFZ 20/56 mg/m² | P1B MM: CFZ 20/70 mg/m² | P1B NHL: CFZ 20/56 mg/m² | P1B NHL: CFZ 20/70 mg/m² | P1B WM: CFZ 20/56 mg/m² | P1B WM: CFZ 20/70 mg/m² | P1B MM: CFZ 20/45 mg/m² + Dex | P1B MM: CFZ 20/56 mg/m² + Dex
Number analyzed (Participants) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 12 | 1 | 0 | 0 | 1 | 4 | 9 | 3
months |  |  | 6.2 [NA to NA] — Not estimable due to the low number of progression events |  |  |  |  |  |  | 9.3 [3.9 to 14.7] | 5.5 [NA to NA] — Could not be calculated since there was only 1 participant with a response | 8.0 [4.1 to 32.5] | 14.8 [NA to NA] — Could not be calculated since there was only 1 participant with a response |  |  | NA [NA to NA] — Not estimable due to the low number of progression events | NA [NA to NA] — Not estimable due to the low number of progression events | 9.0 [1.9 to NA] — Not estimable due to the low number of progression events | 22.6 [17.5 to 27.6]

5. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival (PFS) is the time from start of treatment to disease progression or death (due to any cause), whichever occurred first.
Time Frame: as for outcome 3
Population: Safety population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | P1B ST: CFZ 20 mg/m² Bolus | P1B ST: CFZ 20/27 mg/m² Bolus | P1B ST: CFZ 20/36 mg/m² Bolus | P2 ST: CFZ 20/36 mg/m² Bolus | P1B ST: CFZ 36 mg/m² | P1B ST: CFZ 45 mg/m² | P1B ST: CFZ 20/45 mg/m² | P1B ST: CFZ 20/56 mg/m² | P1B ST: CFZ 20/70 mg/m² | P1B MM: CFZ 20/36 mg/m² | P1B MM: CFZ 20/45 mg/m² | P1b MM: CFZ 20/56 mg/m² | P1B MM: CFZ 20/70 mg/m² | P1B NHL: CFZ 20/56 mg/m² | P1B NHL: CFZ 20/70 mg/m² | P1B WM: CFZ 20/56 mg/m² | P1B WM: CFZ 20/70 mg/m² | P1B MM: CFZ 20/45 mg/m² + Dex | P1B MM: CFZ 20/56 mg/m² + Dex
Number analyzed (Participants) | 3 | 4 | 7 | 65 | 6 | 7 | 6 | 10 | 11 | 4 | 3 | 24 | 2 | 2 | 3 | 1 | 4 | 14 | 8
months | 5.1 [NA to NA] — Could not be estimated due to the low number of events | 1.8 [1.6 to 1.9] | 1.8 [1.0 to NA] — Could not be estimated due to the low number of events | 1.8 [1.7 to 2.1] | 1.7 [1.1 to NA] — Could not be estimated due to the low number of events | 2.9 [0.9 to 15.4] | 1.4 [0.3 to 24.6] | 1.5 [0.3 to 2.0] | 1.6 [0.4 to 5.4] | 5.2 [4.4 to 15.1] | 4.6 [1.4 to 5.9] | 6.9 [1.2 to 8.4] | 9.4 [1.9 to 16.8] | NA [1.6 to NA] — Could not be estimated due to the low number of events | 1.0 [0.6 to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events | 4.6 [1.9 to 12.7] | 11.5 [1.8 to 28.0]

6. Secondary Outcome: Time to Progression
Description: Time to Progression (TTP) is defined as number of months between start of treatment and first evidence/documentation of disease progression.
Time Frame: as for outcome 3
Population: Safety population.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- P1B WM: CFZ 20/70 mg/m²: Participants with Waldenstrom macroglobulinemia (WM) received carfilzomib 20 mg/m² administered by intravenous infusion over 30 minutes on Cycle 1 Days 1 and 2 only, then 56 mg/m² on Days 8, 9, 15 and 16 and thereafter for the remainder of treatment. All participants with stable disease or better after 2 cycles could continue treatment until progressive disease or unacceptable toxicity.
Arm/Group | P1B ST: CFZ 20 mg/m² Bolus | P1B ST: CFZ 20/27 mg/m² Bolus | P1B ST: CFZ 20/36 mg/m² Bolus | P2 ST: CFZ 20/36 mg/m² Bolus | P1B ST: CFZ 36 mg/m² | P1B ST: CFZ 45 mg/m² | P1B ST: CFZ 20/45 mg/m² | P1B ST: CFZ 20/56 mg/m² | P1B ST: CFZ 20/70 mg/m² | P1B MM: CFZ 20/36 mg/m² | P1B MM: CFZ 20/45 mg/m² | P1b MM: CFZ 20/56 mg/m² | P1B MM: CFZ 20/70 mg/m² | P1B NHL: CFZ 20/56 mg/m² | P1B NHL: CFZ 20/70 mg/m² | P1B WM: CFZ 20/56 mg/m² | P1B WM: CFZ 20/70 mg/m² | P1B MM: CFZ 20/45 mg/m² + Dex | P1B MM: CFZ 20/56 mg/m² + Dex
Number analyzed (Participants) | 3 | 4 | 7 | 65 | 6 | 7 | 6 | 10 | 11 | 4 | 3 | 24 | 2 | 2 | 3 | 1 | 4 | 14 | 8
months | 5.1 [NA to NA] — Could not be estimated due to the low number of events | 1.8 [1.6 to 1.9] | 1.8 [1.6 to NA] — Could not be estimated due to the low number of events | 1.8 [1.7 to 2.1] | 1.7 [1.1 to NA] — Could not be estimated due to the low number of events | 1.6 [0.9 to 4.1] | 1.6 [1.1 to NA] — Could not be estimated due to the low number of events | 1.6 [0.5 to 2.0] | 1.6 [0.3 to 5.6] | 5.2 [4.4 to 15.1] | 4.6 [1.4 to 5.9] | 6.9 [1.2 to 8.4] | 9.4 [1.9 to 16.8] | NA [1.6 to NA] — Could not be estimated due to the low number of events | 1.0 [0.6 to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events | 4.6 [1.9 to 12.7] | 11.5 [1.8 to 28.0]

7. Secondary Outcome: Maximum Observed Plasma Concentration of Carfilzomib
Description: Plasma concentrations of carfilzomib were determined by a validated liquid chromatography tandem mass spectrometry method. Concentration values that were below the lower limit of quantification of 0.1 ng/mL were set to zero. Treatment groups receiving the same dose (e.g. 20 mg/m²) were combined for Day 1 analyses.
Time Frame: Cycle 1, Day 1, predose and at 5 minutes and 15 minutes post start of infusion (for 30-minute infusion groups only), and at the end of infusion, 5, 15, and 30 minutes; and 1, 2, and 4 hours after the end of the infusion.
Population: Safety population with available pharmacokinetic (PK) data. PK analyses were conducted in solid tumor and multiple myeloma groups only and were not conducted for lymphoma or participants enrolled under Amendment 4 (CFX + dexamethasone).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- ST: CFZ 20 mg/m² Bolus: Participants with solid tumors received carfilzomib 20 mg/m² administered by bolus intravenous infusion over 2-10 minutes on Cycle 1 Day 1.
- ST: CFZ 20 mg/m²: Participants with solid tumors received carfilzomib 20 mg/m² administered by intravenous infusion over 30 minutes on Cycle 1 Day 1.
- ST: CFZ 36 mg/m²: Participants with solid tumors received carfilzomib 36 mg/m² administered by intravenous infusion over 30 minutes on Day 1.
- ST: CFZ 45 mg/m²: Participants with solid tumors received carfilzomib 45 mg/m² administered by intravenous infusion over 30 minutes on Day 1.
- MM: CFZ 20 mg/m²: Participants with multiple myeloma received carfilzomib 20 mg/m² administered by intravenous infusion over 30 minutes on Cycle 1 Day 1.
Arm/Group | ST: CFZ 20 mg/m² Bolus | ST: CFZ 20 mg/m² | ST: CFZ 36 mg/m² | ST: CFZ 45 mg/m² | MM: CFZ 20 mg/m²
Number analyzed (Participants) | 30 | 21 | 6 | 6 | 30
ng/mL | 2390 (104) | 914 (58.2) | 1061 (50.7) | 1193 (197.3) | 722 (62.1)

8. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of Carfilzomib
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | ST: CFZ 20 mg/m² Bolus | ST: CFZ 20 mg/m² | ST: CFZ 36 mg/m² | ST: CFZ 45 mg/m² | MM: CFZ 20 mg/m²
Number analyzed (Participants) | 30 | 21 | 6 | 6 | 30
hours | 0.0500 [0 to 0.167] | 0.500 [0.0833 to 0.7500] | 0.258 [0.0833 to 0.500] | 0.275 [0.100 to 0.550] | 0.250 [0.0833 to 0.750]

9. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Concentration Measured (AUC0-last) for Carfilzomib
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | ST: CFZ 20 mg/m² Bolus | ST: CFZ 20 mg/m² | ST: CFZ 36 mg/m² | ST: CFZ 45 mg/m² | MM: CFZ 20 mg/m²
Number analyzed (Participants) | 30 | 21 | 6 | 6 | 30
h*ng/mL | 251 (92.0) | 346 (57.4) | 426 (70.1) | 536 (150.4) | 269 (54.3)

10. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC0-inf) for Carfilzomib
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | ST: CFZ 20 mg/m² Bolus | ST: CFZ 20 mg/m² | ST: CFZ 36 mg/m² | ST: CFZ 45 mg/m² | MM: CFZ 20 mg/m²
Number analyzed (Participants) | 23 | 18 | 6 | 6 | 28
h*ng/mL | 223 (104) | 324 (52.8) | 426 (70.1) | 538 (150.1) | 273 (55.3)

11. Secondary Outcome: Elimination Half-life (t½) of Carfilzomib
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | ST: CFZ 20 mg/m² Bolus | ST: CFZ 20 mg/m² | ST: CFZ 36 mg/m² | ST: CFZ 45 mg/m² | MM: CFZ 20 mg/m²
Number analyzed (Participants) | 23 | 18 | 6 | 6 | 28
hours | 0.444 [0.152 to 2.20] | 0.888 [0.368 to 2.33] | 0.917 [0.359 to 1.23] | 0.952 [0.810 to 2.11] | 0.888 [0.411 to 1.57]

12. Secondary Outcome: Clearance (CL) of Carfilzomib
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: liters/hour
Arm/Group | ST: CFZ 20 mg/m² Bolus | ST: CFZ 20 mg/m² | ST: CFZ 36 mg/m² | ST: CFZ 45 mg/m² | MM: CFZ 20 mg/m²
Number analyzed (Participants) | 23 | 18 | 6 | 6 | 28
liters/hour | 263 (398) | 139 (70.1) | 182 (88.8) | 302 (438) | 164 (89.6)

13. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Carfilzomib
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | ST: CFZ 20 mg/m² Bolus | ST: CFZ 20 mg/m² | ST: CFZ 36 mg/m² | ST: CFZ 45 mg/m² | MM: CFZ 20 mg/m²
Number analyzed (Participants) | 23 | 18 | 6 | 6 | 27
liters | 27.7 (48.6) | 31.0 (21.9) | 22.7 (24.2) | 113 (230) | 21.8 (24.6)

14. Secondary Outcome: Mean Residence Time (MRT) Extrapolated to Infinity for Carfilzomib
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ST: CFZ 20 mg/m² Bolus | ST: CFZ 20 mg/m² | ST: CFZ 36 mg/m² | ST: CFZ 45 mg/m² | MM: CFZ 20 mg/m²
Number analyzed (Participants) | 23 | 18 | 6 | 6 | 27
hours | 0.0902 (0.0319) | 0.227 (0.150) | 0.116 (0.0828) | 0.205 (0.156) | 0.117 (0.0799)

ADVERSE EVENTS:
Time Frame: From the first administration of carfilzomib and within 30 days after the last dose of study treatment; maximum duration of treatment was 366 days for bolus administration and 1073 days for infusion
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
  Summary of Adverse Events includes only those subjects who received at least one dose of investigational product.
Arm/Group | P1B ST: CFZ 20 mg/m² Bolus | P1B ST: CFZ 20/27 mg/m² Bolus | P1B ST: CFZ 20/36 mg/m² Bolus | P2 ST: CFZ 20/36 mg/m² Bolus | P1B ST: CFZ 36 mg/m² | P1B ST: CFZ 45 mg/m² | P1B ST: CFZ 20/45 mg/m² | P1B ST: CFZ 20/56 mg/m² | P1B ST: CFZ 20/70 mg/m² | P1B MM: CFZ 20/36 mg/m² | P1B MM: CFZ 20/45 mg/m² | P1B MM: CFZ 20/56 mg/m² | P1B MM: CFZ 20/70 mg/m² | P1B LYM: CFZ 20/56 mg/m² | P1B LYM: CFZ 20/70 mg/m² | P1B MM: CFZ 20/45 mg/m² + Dex | P1B MM: CFZ 20/56 mg/m² + Dex
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/4 | 4/7 | 27/65 | 2/6 | 4/7 | 5/6 | 5/10 | 6/11 | 2/4 | 0/3 | 11/24 | 2/2 | 1/3 | 5/7 | 5/14 | 3/8
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 7/7 | 65/65 | 6/6 | 7/7 | 6/6 | 10/10 | 11/11 | 4/4 | 3/3 | 24/24 | 2/2 | 3/3 | 7/7 | 14/14 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | P1B ST: CFZ 20 mg/m² Bolus (N=3) | P1B ST: CFZ 20/27 mg/m² Bolus (N=4) | P1B ST: CFZ 20/36 mg/m² Bolus (N=7) | P2 ST: CFZ 20/36 mg/m² Bolus (N=65) | P1B ST: CFZ 36 mg/m² (N=6) | P1B ST: CFZ 45 mg/m² (N=7) | P1B ST: CFZ 20/45 mg/m² (N=6) | P1B ST: CFZ 20/56 mg/m² (N=10) | P1B ST: CFZ 20/70 mg/m² (N=11) | P1B MM: CFZ 20/36 mg/m² (N=4) | P1B MM: CFZ 20/45 mg/m² (N=3) | P1B MM: CFZ 20/56 mg/m² (N=24) | P1B MM: CFZ 20/70 mg/m² (N=2) | P1B LYM: CFZ 20/56 mg/m² (N=3) | P1B LYM: CFZ 20/70 mg/m² (N=7) | P1B MM: CFZ 20/45 mg/m² + Dex (N=14) | P1B MM: CFZ 20/56 mg/m² + Dex (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 5 | 0 | 0 | 2 | 1 | 4 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatorenal failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 1
Rhinovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour lysis syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuritis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Visual field defect (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Laryngeal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | P1B ST: CFZ 20 mg/m² Bolus (N=3) | P1B ST: CFZ 20/27 mg/m² Bolus (N=4) | P1B ST: CFZ 20/36 mg/m² Bolus (N=7) | P2 ST: CFZ 20/36 mg/m² Bolus (N=65) | P1B ST: CFZ 36 mg/m² (N=6) | P1B ST: CFZ 45 mg/m² (N=7) | P1B ST: CFZ 20/45 mg/m² (N=6) | P1B ST: CFZ 20/56 mg/m² (N=10) | P1B ST: CFZ 20/70 mg/m² (N=11) | P1B MM: CFZ 20/36 mg/m² (N=4) | P1B MM: CFZ 20/45 mg/m² (N=3) | P1B MM: CFZ 20/56 mg/m² (N=24) | P1B MM: CFZ 20/70 mg/m² (N=2) | P1B LYM: CFZ 20/56 mg/m² (N=3) | P1B LYM: CFZ 20/70 mg/m² (N=7) | P1B MM: CFZ 20/45 mg/m² + Dex (N=14) | P1B MM: CFZ 20/56 mg/m² + Dex (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 17 | 1 | 1 | 2 | 4 | 3 | 2 | 1 | 10 | 1 | 1 | 2 | 5 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 3 | 10 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 1 | 1 | 3 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 3 | 1 | 1 | 13 | 2 | 1 | 3 | 5 | 3
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenopia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Visual disturbance (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 12 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 14 | 0 | 1 | 2 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 1 | 11 | 0 | 2 | 2 | 4 | 3 | 1 | 0 | 2 | 0 | 0 | 1 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | 18 | 1 | 1 | 2 | 2 | 1 | 0 | 1 | 6 | 1 | 1 | 3 | 1 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 8 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Faeces pale (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Gastric outlet obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Gingival swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 4 | 28 | 2 | 4 | 2 | 4 | 6 | 3 | 2 | 13 | 1 | 1 | 1 | 4 | 3
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral soft tissue disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomach discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 4 | 18 | 2 | 4 | 2 | 1 | 3 | 2 | 1 | 8 | 1 | 1 | 1 | 4 | 0
Asthenia (General disorders) | 0 | 0 | 4 | 7 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 1 | 2
Axillary pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breakthrough pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Catheter related complication (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 5 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 2 | 18 | 1 | 1 | 3 | 2 | 2 | 1 | 2 | 8 | 0 | 0 | 4 | 0 | 1
Difficulty in walking (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 3 | 38 | 0 | 4 | 3 | 4 | 5 | 3 | 3 | 14 | 2 | 2 | 3 | 9 | 5
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Implant site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion site erythema (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion site pain (General disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Infusion site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Irritability (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Malaise (General disorders) | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 2 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 2 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 9 | 0 | 0 | 2 | 3 | 1 | 2 | 1 | 5 | 0 | 1 | 1 | 3 | 1
Pain (General disorders) | 0 | 0 | 0 | 7 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 3 | 17 | 1 | 1 | 2 | 5 | 2 | 1 | 1 | 13 | 1 | 3 | 5 | 2 | 4
Temperature intolerance (General disorders) | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thirst (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Multiple allergies (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dental caries (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungaemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal rash (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 1 | 1 | 0 | 2
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 5 | 1 | 0 | 3 | 7 | 4
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 5 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contrast media reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 7 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeding tube complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Incision site complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 11 | 0 | 3 | 1 | 3 | 2 | 0 | 2 | 6 | 0 | 0 | 4 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Blood pressure orthostatic decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Creatinine renal clearance decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Heart rate increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza serology positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Methicillin-resistant staphylococcal aureus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 26 | 0 | 2 | 1 | 0 | 2 | 2 | 0 | 4 | 0 | 0 | 0 | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 9 | 0 | 2 | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 3 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 3 | 8 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 5 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 4 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 10 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 5 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 15 | 0 | 1 | 2 | 3 | 1 | 1 | 0 | 4 | 0 | 0 | 1 | 3 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 5 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 7 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 5 | 1 | 1 | 2 | 3 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 5 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 7 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 1 | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 8 | 0 | 2 | 0 | 2 | 0 | 1 | 1 | 3 | 0 | 1 | 0 | 5 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 6 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Areflexia (Nervous system disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Coordination abnormal (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 10 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 7 | 0 | 2 | 1 | 3 | 1
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 9 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 4 | 13 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 8 | 1 | 1 | 1 | 5 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 11 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyporeflexia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neuropathic pain (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 3 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 6 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Speech disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 9 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 4 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 3 | 9 | 0 | 2 | 0 | 3 | 1 | 0 | 1 | 7 | 0 | 0 | 2 | 5 | 3
Mood altered (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neurogenic bladder (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 3 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine flow decreased (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 12 | 0 | 1 | 2 | 2 | 2 | 1 | 1 | 7 | 1 | 2 | 3 | 8 | 2
Crackles lung (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 23 | 2 | 2 | 1 | 2 | 3 | 1 | 0 | 12 | 0 | 2 | 3 | 6 | 2
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 5 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 3 | 1 | 0 | 1 | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 5 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 5 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 4 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 2
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 5 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Leukoplakia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 10 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 6 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin tightness (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 5 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 9 | 1 | 1 | 1 | 6 | 2
Hypotension (Vascular disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.